CLINICAL TRIAL: NCT06293794
Title: New Solutions to Support Evidence-based Prescribing for Heart Failure
Brief Title: Decision Support for Heart Failure Prescribing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0991
Record Dates: First submitted 2024-02-06; First posted 2024-03-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Decision Support Systems, Clinical; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Compare traditional and personalized CDS in a pragmatic randomized controlled trial at one health system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Clinical Decision Support (CDS) (Experimental)
  Interventions: Other: Traditional Clinical Decision Support (CDS)
- Personalized Clinical Decision Support (CDS) (Experimental)
  Interventions: Other: Personalized Clinical Decision Support (CDS)

INTERVENTIONS:
Other: Personalized Clinical Decision Support (CDS) — The personalized CDS intervention evaluates clinician past prescribing patterns to determine whether prescribing misconceptions might exist and then conditionally present information to address those misconceptions. This is done through a nudge in the electronic health record that addresses common prescribing misconceptions for heart failure.
  Arms: Personalized Clinical Decision Support (CDS)
Other: Traditional Clinical Decision Support (CDS) — The traditional CDS is the usual care intervention, which is patient-specific but are not clinician-specific.
  Arms: Traditional Clinical Decision Support (CDS)

SUMMARY:
Clinical decision support (CDS) tools can 'nudge' clinicians to make the best decisions easy. Although required by "meaningful use" regulations, more than 40% of CDS lead to no change and the remaining lead to improvements that are modest at best. This is because CDS tools often ignore contextual factors and present irrelevant information. Although many tools have undergone patient-specific optimization, 'traditional CDS' are rarely clinician-specific. For example, a traditional CDS tool for beta blockers and heart failure with reduced ejection fraction (HFrEF) addresses common prescribing misconceptions by stating asthma is not a contraindication and providing a safe threshold for blood pressure. For clinicians without these misconceptions, these statements are irrelevant and distract from key information. A 'personalized CDS' would evaluate clinician past prescribing patterns to determine whether prescribing misconceptions might exist and then conditionally present information to address those misconceptions. The objective of this research is to create personalized clinician-specific CDS that overcome shortcomings of traditional CDS. The central hypothesis is a personalized CDS that minimizes irrelevant information will lead to a higher rate of prescribing guideline-directed management and therapy (GDMT) for HFrEF compared to a traditional CDS.

ELIGIBILITY:
Inclusion Criteria:

* The study subjects are potential users of the CDS, specifically clinicians with prescribing privileges who practice at one of the health system's (UCHealth) outpatient cardiology or primary care clinics. Because we are observing their prescribing behaviors, we are also evaluating patient characteristics which could influence their prescribing decisions.

Exclusion Criteria:

* Clinicians who do not practice in cardiology or primary care clinics or do not practice within UCHealth system.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of CDS alerts resulting in the prescription of a recommended medication | 6 months
  The primary outcome is number of CDS alerts that resulted in the prescription of the medication recommended by the CDS alert. Recommended medications include either evidence-based beta blockers, sacubitril/valsartan, mineralocorticoid receptor antagonists or sodium/glucose cotransport 2 inhibitors. Prescriptions will be based on actual prescription orders instead of clinician-stated responses, given the latter may overestimate effectiveness.

SECONDARY OUTCOMES:
Number of patients the CDS alerted for | 6 months
  This outcome evaluates the reach of the CDS by counting the number of patients that the CDS alerted for.
Number of alerts that were not outright dismissed | 6 months
  This outcome will help investigators understand if the CDS id being used or dismissed.
Number of prescription orders for guideline directed management and therapies (GDMT) for heart failure | 6 months
  This outcome measures the number of prescriptions for each of the four categories of GDMT: evidence-based beta blockers, sacubitril/valsartan, mineralocorticoid receptor antagonists or sodium/glucose cotransport 2 inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Katy E Trinkley, PharmD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCHealth Primary Care and Cardiology Outpatient Clinics, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in related areas of interest. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (e.g., data use/sharing agreements) are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in related areas of interest. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (e.g., data use/sharing agreements) are prerequisites to the sharing of data with the requesting party. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement.